CLINICAL TRIAL: NCT04512183
Title: Effectiveness of Simulation in the Cognitive, Physiological and Emotional Sphere of Nursing Students in Caring for Patients With Signs of Sepsis: Crossover Clinical Trial
Brief Title: Effectiveness of Simulation With Nursing Students in the Care of Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcia Cristina da Silva Magro, Principal Investigator; PhD, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 3906816
Record Dates: First submitted 2020-08-02; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Learning Process in Nursing Graduation; Stress
Keywords: Simulation; Stress, Psychological; Nursing, Education; Simulation Training; Learning
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Fidelity Simulation (Experimental): First, students will go through an inverted class on sepsis. Then, they will be submitted to high-fidelity simulation scenarios to care for patients with sespe. After the scenario, the students' physiological parameters (blood pressure, heart rate, body temperature, respiratory rate and oxygen saturation) will be measured. After the scenario, students will go through a reflective debriefing session.
  Interventions: Other: High-Fidelity Simulation
- Low-Fidelity Simulation (Active Comparator): First, students will go through an inverted class on sepsis. Then, they will be submitted to low-fidelity simulation scenarios to care for patients with sespe. After the scenario, the students' physiological parameters (blood pressure, heart rate, body temperature, respiratory rate and oxygen saturation) will be measured. After the scenario, students will go through a feedback session.
  Interventions: Other: Low-Fidelity Simulation

INTERVENTIONS:
Other: High-Fidelity Simulation — Teaching strategy based on high-fidelity simulation, which simulates the reality of health care to promote meaningful learning.
  Arms: High-Fidelity Simulation
Other: Low-Fidelity Simulation — Teaching strategy based on low-fidelity simulation, which simulates the reality of health care using less technological and less interactive mannequins.
  Arms: Low-Fidelity Simulation

SUMMARY:
Simulation is an active teaching strategy capable of reproducing real situations and allowing practical experiences, in which the student is the protagonist of his own knowledge. Scientific evidence highlights, that exposure to the unknown or new can generate stress to the individual, but when dosed, to a certain extent it can increase the level of knowledge. Not infrequently, the lack of stress control can trigger physiological and subjective changes resulting from the increase in its level, such as situations that include the implementation of simulation scenarios in pedagogical teaching models.

DETAILED DESCRIPTION:
Objective:

To evaluate the effect of simulation (high and low fidelity) on the cognitive, physiological and emotional sphere of nursing students in caring for patients with signs of sepsis.

Hypothesis of the study:

Null hypothesis: Students undergoing high-fidelity simulation will show similar levels of stress, cognitive performance and retention of knowledge in relation to those who will perform low-fidelity simulation in patients with signs of sepsis.

Alternative hypothesis: The cognitive performance and stress will be higher in students who experience high fidelity simulation when compared to students who experience low fidelity simulation.

ELIGIBILITY:
Inclusion Criteria:

* Students approved in the discipline related to nursing care for adult and elderly patients;
* Aged over 18 years.

Exclusion Criteria:

* Who have experience in the health field (firefighters and nursing technicians, among others);
* Members of the Health Simulation League;
* Those who do not complete all stages of the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Performance (Baseline) | Applied before the intervention
  Students' knowledge about nursing care in sepsis measured using a structured questionnaire with six multiple-choice questions
Cognitive Performance (Post-test) | Applied immediately after the intervention
  Students' knowledge about nursing care in sepsis measured using a structured questionnaire with six multiple-choice questions
Cognitive Performance (Retention) | Applied thirty days after the intervention
  Students' knowledge about nursing care in sepsis measured using a structured questionnaire with six multiple-choice questions

SECONDARY OUTCOMES:
Student stress (Baseline) | Before the intervention
  Assessment of students' stress intensity with pedagogical activities through the application of the Kezkak Stress Scale. This scale has 31 items of the Likert type of 4 points, being: 1 - Nothing stressful; 2 - A little stressful; 3 - Very stressful; 4 - Extremely stressful. The value 1 means less stress and 4 more stress.
Student stress (Post-test) | Immediately after the intervention
  Assessment of students' stress intensity with pedagogical activities through the application of the Kezkak Stress Scale. This scale has 31 items of the Likert type of 4 points, being: 1 - Nothing stressful; 2 - A little stressful; 3 - Very stressful; 4 - Extremely stressful. The value 1 means less stress and 4 more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia CS Magro, PhD, Principal Investigator — University of Brasilia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boostel R, Felix JVC, Bortolato-Major C, Pedrolo E, Vayego SA, Mantovani MF. Stress of nursing students in clinical simulation: a randomized clinical trial. Rev Bras Enferm. 2018 May;71(3):967-974. doi: 10.1590/0034-7167-2017-0187. English, Portuguese. PMID 29924167
- [Background] Kaneko RMU, Lopes MHBM. Realistic health care simulation scenario: what is relevant for its design? Rev Esc Enferm USP. 2019 May 30;53:e03453. doi: 10.1590/S1980-220X2018015703453. English, Portuguese. PMID 31166535
- [Background] Bingham AL, Sen S, Finn LA, Cawley MJ. Retention of advanced cardiac life support knowledge and skills following high-fidelity mannequin simulation training. Am J Pharm Educ. 2015 Feb 17;79(1):12. doi: 10.5688/ajpe79112. PMID 25741028
- [Background] Machado FR, Assuncao MS, Cavalcanti AB, Japiassu AM, Azevedo LC, Oliveira MC. Getting a consensus: advantages and disadvantages of Sepsis 3 in the context of middle-income settings. Rev Bras Ter Intensiva. 2016 Oct-Dec;28(4):361-365. doi: 10.5935/0103-507X.20160068. No abstract available. PMID 28099632
- [Background] Englert NC, McDermott D. Back to Fundamentals: Using High- and Low-Fidelity Simulation to Provide Reinforcement of Preventative Measures for Sepsis. Crit Care Nurs Q. 2016 Jan-Mar;39(1):14-23. doi: 10.1097/CNQ.0000000000000097. PMID 26633154